CLINICAL TRIAL: NCT05171361
Title: Pancreaticogastrostomy Versus Pancreaticojejunostomy With Dunking Technique After Pancreaticodudenectomy: A Prospective Randomized Comparative Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherif Alaa, resident doctor, Assiut University
Other Study IDs: Pancreaticojejunostomy
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Pancreaticobiliary Cancer
Keywords: pancreaticojejunostomy; pancreaticogastrostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreaticojejunostomy: With Dunking Technique after Pancreaticodudenectomy
  Interventions: Procedure: Pancreaticogastrostomy versus Pancreaticojejunostomy with Dunking Technique
- Pancreaticogastrostomy: With Dunking Technique after Pancreaticodudenectomy
  Interventions: Procedure: Pancreaticogastrostomy versus Pancreaticojejunostomy with Dunking Technique

INTERVENTIONS:
Procedure: Pancreaticogastrostomy versus Pancreaticojejunostomy with Dunking Technique — To compare between the outcomes of pancreaticogastrostomy and pancreaticojejunostomy with dunking technique after Pancreaticodudenectomy

SUMMARY:
To compare between the outcomes of pancreaticogastrostomy and pancreaticojejunostomy with dunking technique after Pancreaticodudenectomy in the treatment of operable periampullary malignancies.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy remains the treatment of choice for periampullary malignancies. Advances in pancreatic surgery techniques and perioperative care have led to reduced mortality rates for Pancreaticodudenectomy [1]. However, morbidity after pancreatic resection remains high, with 30-60% of patients experiencing complications following surgery, mainly as a result of leak and subsequent fistula from the pancreatic anastomosis [2].The leakage of the pancreatic anastomosis remains the most serious problem as it is the major cause of morbidity after pancreaticoduodenectomy, and also contributes significantly to prolonged hospitalization [5]. For this reason, surgeons have always directed their efforts at reducing the rate of pancreatic fistula through the introduction of new and effective methods of construction of the pancreatic anastomosis [6]. Various techniques have been described for joining the pancreatic stump either with the jejunum or with the stomach, with or without internal or external drainage of the pancreatic duct. Recently, new prospective randomized studies have demonstrated the advantage of pancreaticogastrostomy over pancreaticojejunostomy in reducing the incidence of pancreatic fistula [3]; however, none of these techniques has proved to be superior in minimizing postoperative mortality and morbidity [4]. One of the difficulties of pancreatic reconstruction after pancreaticoduodenectomy is the presence of soft pancreas which leads to high risk of fistula so dunking technique was raised [8]. But few researches or papers have focused on its efficacy and even fewer papers have discussed dunking in pancreaticogastrostomy and pancreaticojejunostomy, So this is the interest of our study to compare between the efficacies of these two techniques.

ELIGIBILITY:
Inclusion Criteria:

* All cases of resectable periampullary carcinomas (cancer head of pancreas, ampullary carcinoma, distal cholangiocarcinoma and second part of duodenum adenocarcinoma) that are surgically fit according to ASA.

Exclusion Criteria:

* 1. Surgically unfit cases according to ASA 2. Locally advanced irresectable cases
* Abutment or encasement of coeliac trunk
* Encasement of SMA less than 180 degree of its axis
* Encasement of portal/SMV more than 180 degree of its axis or infiltration segment too long more than 2.5 cm that the remaining segment will not coapts after resection.

  3. Metastatic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases of resectable periampullary carcinomas
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative anastomosis leakage | One month
  Compare between dunking in pancreaticogastrostomy and pancreaticojejunostomy and the rate of postoperative anastomosis leakage

REFERENCES:
- [Background] Cheng Y, Briarava M, Lai M, Wang X, Tu B, Cheng N, Gong J, Yuan Y, Pilati P, Mocellin S. Pancreaticojejunostomy versus pancreaticogastrostomy reconstruction for the prevention of postoperative pancreatic fistula following pancreaticoduodenectomy. Cochrane Database Syst Rev. 2017 Sep 12;9(9):CD012257. doi: 10.1002/14651858.CD012257.pub2. PMID 28898386
- [Background] Que W, Fang H, Yan B, Li J, Guo W, Zhai W, Zhang S. Pancreaticogastrostomy versus pancreaticojejunostomy after pancreaticoduodenectomy: a meta-analysis of randomized controlled trials. Am J Surg. 2015 Jun;209(6):1074-82. doi: 10.1016/j.amjsurg.2014.07.019. Epub 2015 Jan 22. PMID 25743406